CLINICAL TRIAL: NCT02432599
Title: Interest of the F18-choline as a Second Line of the Tracer for Detection of Parathyroid Adenomas
Acronym: APACH1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APACH1
Record Dates: First submitted 2015-04-29; First posted 2015-05-04 (Estimated); Last update posted 2018-01-04 (Actual); Status verified 2016-08

CONDITIONS: Hyperparathyroidism
Keywords: F18-choline
MeSH Terms: conditions — Hyperparathyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- F18-choline PET (Experimental): F18-choline PET examination will be performed before surgery
  Interventions: Radiation: F18-choline PET examination

INTERVENTIONS:
Radiation: F18-choline PET examination — F18-choline PET examination will be performed before surgery

SUMMARY:
The rationale for the proposed pilot study is to investigate the ability of PET-CT with F18-choline to detect and locate the parathyroid adenoma in patients with primary hyperparathyroidism and negative or non-contributory MIBI (Tc-99m sestamibi) and cervical ultrasound, in order to avoid unnecessary bilateral cervical exploration.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years or more;
* Patient with a primary hyperparathyroidism and witj a negative or non-contriburatory MIBI parathyroid scintigraphy and neck ultrasonography, for which surgical resection is planned;
* Confirmation of the diagnosis of primary hyperparathyroidism on laboratory tests
* Affiliate to a social security system;
* Patient written informed consent.

Exclusion Criteria:

* Patient deprived of liberty, under guardianship;
* Any medical or psychological condition witch could compromise the capacity of the patient to participate in the study;
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2015-03; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity (ability to identify and visualize the parathyroid adenoma) | Up to 2 months
  Sensitivity of PET-CT with F18-choline (FCH) to identify and visualize the parathyroid adenoma in patients with primary hyperparathyroidism and negative or non-contributory parathyroid scintigraphy MIBI and cervical ultrasound

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU, Caen
  - Centre François Baclesse, Caen

REFERENCES:
- [Derived] Quak E, Blanchard D, Houdu B, Le Roux Y, Ciappuccini R, Lireux B, de Raucourt D, Grellard JM, Licaj I, Bardet S, Reznik Y, Clarisse B, Aide N. F18-choline PET/CT guided surgery in primary hyperparathyroidism when ultrasound and MIBI SPECT/CT are negative or inconclusive: the APACH1 study. Eur J Nucl Med Mol Imaging. 2018 Apr;45(4):658-666. doi: 10.1007/s00259-017-3911-1. Epub 2017 Dec 22. PMID 29270788